CLINICAL TRIAL: NCT01246102
Title: Phase I Study of the HSP-90 Inhibitor, AT13387, in Adults With Refractory Solid Tumors
Brief Title: AT13387 in Adults With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110029; 11-C-0029; NCT01245218 (obsolete NCT alias)
Record Dates: First submitted 2010-11-20; First posted 2010-11-23 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2017-10-27

CONDITIONS: Solid Tumors; Breast Cancer
Keywords: Targeted Therapy; HER2 Positive Cancer; Cancer; Solid Tumor; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — (2,4-dihydroxy-5-isopropylphenyl)-(5-(4-methylpiperazin-1-ylmethyl)-1,3-dihydroisoindol-2-yl)methanone

ARMS (1):
- 1 (Experimental): starting at 20 mg/m2
  Interventions: Drug: AT13387

INTERVENTIONS:
Drug: AT13387 — Treatment will be administered as a 1-hour IV infusion on 2 consecutive days of every week for 3 weeks, followed by a 1-week period without drug administration.

SUMMARY:
Background:

- The experimental drug AT13387 has been shown to have some anticancer effects against tumor cells by blocking a protein that affects other proteins inside certain cancer cells, and helps to prevent the cancer cells from reproducing and spreading. AT13387 has not been tested in humans, and researchers are interested in investigating whether it can be used to treat solid tumors that have not responded to standard treatments.

Objectives:

- To investigate the safety and effectiveness of AT13387 in individuals with solid tumors.

Eligibility:

- Individuals at least 18 years of age who have solid tumors that have not responded to standard treatments.

Design:

* Participants will be screened with a physical examination and medical history, as well as blood tests and tumor imaging studies.
* AT13387 will be given in 28-day cycles of treatment. Participants will receive AT13387 twice a week (2 days in a row) for the first 3 weeks of the cycle, followed by a fourth week without the drug.
* Participants will have regular blood and urine samples, imaging studies, eye examinations, and tumor biopsies to monitor the effects of the treatment.
* Participants will continue treatment with AT13387 unless serious side effects develop or the tumor stops responding to treatment.

DETAILED DESCRIPTION:
Background:

* AT13387 is a synthetic Hsp90 inhibitor that has demonstrated improved characteristics over other Hsp90 inhibitors. AT13387 has a long tumor retention half-life and prolonged inhibitory effect on its known oncogenic client proteins.
* AT13387 has demonstrated activity against multiple cancer cell lines and tumor xenografts in pre-clinical models.

Primary Objectives:

* Define the safety and tolerability of AT13387 administered on a QDx2 every week, 3 weeks out of 4 scheduled, in adults with refractory solid tumors.
* Establish the maximum tolerated dose (MTD) of AT13387 administered on a QDx2 every week, 3 weeks out of 4 schedule, in adults with refractory solid tumors.

Secondary Objectives:

* Determine the pharmacokinetics (PK) of AT13387 administered on a QDx2 every week, 3 weeks out of 4 schedule, in adults with refractory solid tumors.
* Assess pharmacodynamic (PD) markers of Hsp90 inhibition and modulation of Hsp90 client proteins by AT13387 in tumor tissue, serum, and PBMCs.

Eligibility:

-Study participants must have histologically confirmed solid tumor malignancy that has progressed or recurred after at least one line of chemotherapy, or for which no standard treatment option exists. Participants enrolling in the expansion phase must have disease amenable to biopsy with willingness to undergo pre- and post-treatment biopsies (Remove the HER 2 archival tissue).

Study Design:

* This study will follow an accelerated titration design 2B with initial dose levels increased in 100% increments.
* The accelerated phase ends when one patient experiences a dose-limiting toxicity or two patients experience Grade 2 drug-related toxicity during the first cycle; when dose level 3 is reached; or at first instance of Grade 2 ocular toxicity in any cycle.
* AT13387 will be administered intravenously, over 1 hour, on 2 consecutive days, 3 out of 4 weeks, every 28 days (i.e., on days 1, 2, 8, 9, 15, and 16 of each 28-day cycle).
* PK and PD studies will be conducted in cycle 1 only. Once the MTD is established, 10 additional patients, will be entered at the MTD to further define toxicity and perform PD studies at this dose; pre- and post-treatment tumor biopsies will be mandatory for these patients.
* CT scans will be performed at baseline and every 2 cycles for restaging.
* Up to 37 patients may be treated.
* Study participants will be offered optional participation in an ongoing NCI imaging study at baseline with a repeat scan following the last dose of AT13387 in cycle 1.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically documented (confirmed at the Laboratory of Pathology, NCI) solid tumor malignancy that is metastatic or unresectable, for which standard curative measures do not exist, or have failed at least one line of standard therapy.
* Patients must have measurable or evaluable disease.
* Patients must have completed any chemotherapy, radiation therapy, or biologic therapy greater than or equal to 4 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C).

Patients must be greater than or equal to 2 weeks since any prior administration of a study drug in an exploratory IND/Phase 0 study. Patients must have recovered to eligibility levels from prior toxicity or adverse events. Patients receiving bisphosphonates for any cancer are eligible to participate.

* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of AT13387 in patients < 18 years of age, children are excluded from this study.
* The Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Life expectancy > 3 months.
* Patients must have normal or adequate organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,500/microL
  * Platelets greater than or equal to 100,000/microL
  * Total bilirubin less than or equal to 1.5 times institutional ULN
  * AST (SGOT)/ALT (SGPT) less than or equal to 2.5 times institutional ULN
  * Creatinine <1.5 times ULN; OR
  * Measured creatinine greater than or equal to 60 mL/minute for patients with clearance creatinine levels greater than or equal to 1.5 times ULN
* The effects of AT13387 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry, for the duration of study participation, and for 2 months after completion of study. Women of childbearing potential must have a negative pregnancy test within 72 hours of enrollment in order to be eligible. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk to nursing infants secondary to treatment of the mother with AT13387, breastfeeding should be discontinued if the mother is treated with AT13387.
* During the expansion phase of the protocol, patients must have:

  * Disease amenable to biopsy
  * Willingness to undergo pre- and post-treatment biopsies
* Ability to understand and the willingness to sign a written informed consent document.
* Currently enrolling in the expansion phase. Patients must have:
* Disease amenable to biopsy
* Willingness to undergo pre- and post-treatment biopsies

EXCLUSION CRITERIA:

* Patients with known brain metastases or carcinomatous meningitis are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for greater than or equal to 2 months after treatment of the brain metastases, without steroids or anti-seizure medications. These patients may be enrolled at the discretion of the principal investigator.
* Patients with clinically significant intercurrent illnesses, including but not limited to, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* QTc > 450 msec for men and > 470 msec for women.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for PK interactions with AT13387.
* Pregnant women are ineligible because the effects of AT13387 on the developing human fetus are unknown.
* Exclude patients with active gastrointestinal bleeding or an event of gastrointestinal bleeding within a week of starting treatment.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women, and members of all races and ethnic groups, are eligible for this trial.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-11-19; Primary Completion 2013-12-30 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Define the safety and tolerability of AT13387; establishing the MTD of At13387 | 3 weeks

SECONDARY OUTCOMES:
Determine the pharmacokinetics (PK) of AT13387; Assess pharmacodynamic (PD) markers of Hsp90 inhibition and modulation of Hsp90 client proteins by AT13387 | After 1 cycle

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Pick E, Kluger Y, Giltnane JM, Moeder C, Camp RL, Rimm DL, Kluger HM. High HSP90 expression is associated with decreased survival in breast cancer. Cancer Res. 2007 Apr 1;67(7):2932-7. doi: 10.1158/0008-5472.CAN-06-4511. PMID 17409397
- [Background] Whitesell L, Mimnaugh EG, De Costa B, Myers CE, Neckers LM. Inhibition of heat shock protein HSP90-pp60v-src heteroprotein complex formation by benzoquinone ansamycins: essential role for stress proteins in oncogenic transformation. Proc Natl Acad Sci U S A. 1994 Aug 30;91(18):8324-8. doi: 10.1073/pnas.91.18.8324. PMID 8078881
- [Background] Bagatell R, Whitesell L. Altered Hsp90 function in cancer: a unique therapeutic opportunity. Mol Cancer Ther. 2004 Aug;3(8):1021-30. PMID 15299085
- [Derived] Do K, Speranza G, Chang LC, Polley EC, Bishop R, Zhu W, Trepel JB, Lee S, Lee MJ, Kinders RJ, Phillips L, Collins J, Lyons J, Jeong W, Antony R, Chen AP, Neckers L, Doroshow JH, Kummar S. Phase I study of the heat shock protein 90 (Hsp90) inhibitor onalespib (AT13387) administered on a daily for 2 consecutive days per week dosing schedule in patients with advanced solid tumors. Invest New Drugs. 2015 Aug;33(4):921-30. doi: 10.1007/s10637-015-0255-1. Epub 2015 Jun 18. PMID 26082332